CLINICAL TRIAL: NCT04384354
Title: Digestive Events in Duchenne Muscular Dystrophy Patients
Acronym: DIGD
Status: Completed | Type: Observational
Sponsor: Centre d'Investigation Clinique et Technologique 805 (Other)
Responsible Party: Principal Investigator, Crenn, Professor, Centre d'Investigation Clinique et Technologique 805
Other Study IDs: DIGDMD
Record Dates: First submitted 2019-07-19; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Duchenne Muscular Dystrophy
Keywords: pseudo occlusion; gastrostomy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Relation between clinical and genetic features and acute digestive events in Duchenne muscular dystrophy patients

DETAILED DESCRIPTION:
Clinical Data of the disease Digestive events (pseudo occlusion, gastrostomy, cholecystectomy) Nutritionnal parameters Genetic of dystrophin (approved genetic nationnal Data base, CHU Cochin, Paris France)

ELIGIBILITY:
Inclusion Criteria:

* all Duchenne muscular dystrophy patients in our center

Exclusion Criteria:

* none

Min Age: 15 Years | Sex: Male
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only male patients, due to the specific disease (Duchenne muscular dystrophy patients)
Study Population: Duchenne muscular dystrophy patients
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Incidence of digestive events | 11 years
  Clinical parameters (yes or no): gastrostomy, bowel occlusion, acute gastric paresia, biliary complication
Prevalence of digestive events | 11 years
  Clinical parameters (yes or no) : gastrostomy, bowel occlusion, acute gastric paresia, biliary complication
Risk factors for digestive events (1) | 11 years
  age (years)
Risk factors for digestive events (2) | 11 years
  pulmonary functional tests (vital capacity in ml/kg)
Risk factors for digestive events (3) | 11 years
  echocardiography parameters (LVEF: left ventricular ejection fraction in %)
Risk factors for digestive events (4) | 11 years
  residual dystrophin level (Western blot and/or immunohistochemistry in muscle)
Risks factors for digestive events (5) | 11 years
  genetic parameters (type of mutation, functional domain of altered dystrophin)

SECONDARY OUTCOMES:
Nutritional status (1) | 11 years
  Weigh (kg) and height (in m) agregated in BMI (kg/m^2)
Nutritional status (2) | 11 years
  albuminemia in g/L

CONTACTS AND LOCATIONS:
Overall Officials: CICIT805 Garches, Study Chair — APHP/UVSQ
Locations (1):
- CICIT805, Garches, France

IPD SHARING:
Plan to Share IPD: Undecided
All clinician and biologist involved in the follow-up of these patients